CLINICAL TRIAL: NCT01941498
Title: A Prospective, Global, Multi-Center Study for the Evaluation of Outcomes on Subjects Undergoing Myopic Treatments Using the WaveLight® Refractive Suite
Brief Title: WaveLight® Refractive Myopic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A01353
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Results first posted 2015-03-11 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Refractive Error
Keywords: nearsighted; farsighted; astigmatism; LASIK; refractive surgery; WaveLight
MeSH Terms: conditions — Refractive Errors; Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WaveLight Refractive Suite (Experimental): LASIK surgery (laser in situ keratomileusis) per standard of care
  Interventions: Device: Wavelight® Refractive Suite; Procedure: LASIK surgery

INTERVENTIONS:
Device: Wavelight® Refractive Suite — Excimer EX500 and Femtosecond FS200 lasers (Wavelight® Refractive Suite) used during LASIK surgery for corneal flap creation and corneal ablation
Procedure: LASIK surgery — Surgical procedure for treating refractive error based on corneal reshaping

SUMMARY:
The purpose of this study is to evaluate outcomes of subjects undergoing myopic surgery using the WaveLight® Refractive Suite (Excimer EX500 and Femtosecond FS200 lasers).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign an informed consent form.
* Have refractive error (in both eyes) that requires refractive surgery.
* Willing to undergo LASIK surgery using the Wavelight® Refractive Suite.
* Myopia between 0.00 to -12.0 diopters pre-operatively.
* Astigmatism between 0.00 to +6.00 diopters pre-operatively.
* Willing and able to attend post-operative examinations per protocol schedule.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Participation in a clinical study within the last 30 days.
* History of previous corneal surgery in either eye.
* Multifocal ablations in either eye.
* PRK or PTK surgery in either eye.
* Suffering from acute or recurring eye diseases in either eye, such as corneal ulcers, cataract, etc.
* Any ocular disease and/or condition that, in the Investigator's clinical judgment, may put subject at significant risk, compromise study results, or interfere significantly with subject's participation in the study.
* Unable to discontinue contact lens wear as specified in protocol.
* History of Herpes simplex or Herpes zoster keratitis.
* Active ocular rosacea.
* Lyme disease.
* History of dry eye that is unresponsive to treatment.
* Severe ocular allergies.
* Other medical conditions and use of medications as specified in protocol.
* Pregnant or planning to become pregnant during the study.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-09; Primary Completion 2014-01 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, GMA, Surgical, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 2 study centers located in the US, 1 study center located in Ireland, and 1 study center located in Germany.
Pre-assignment Details: Of the 104 enrolled participants, 7 were exited prior to surgery as screen failures. This reporting group includes all enrolled participants who underwent LASIK surgery (97).
Groups:
- WaveLight Refractive Suite: Excimer EX500 and Femtosecond FS200 lasers used during LASIK surgery for corneal flap creation and corneal ablation
Period: Overall Study
Arm/Group | WaveLight Refractive Suite
Started | 97
Completed | 96
Not Completed | 1
Not completed — Relocated out of state | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all enrolled participants.
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Difference in Binocular UCVA at 1 Month Post-Treatment and Pre-Treatment Binocular BCVA
Description: Visual acuity (VA) with corrective devices (BCVA) was assessed binocularly (both eyes together) pre-treatment and subtracted from VA without spectacles or other visual corrective devices (UCVA) assessed binocularly at 1 month post-treatment. VA was measured at a distance of 4 meters and reported in logMAR (logarithm of the minimum angle of resolution), with 0.00 logMAR corresponding to 20/20 Snellen. A negative value indicates an improvement in VA from pre-treatment to Month 1.
Time Frame: Month 1
Population: This analysis population includes all participants with 1 month post-operative measurement of the primary efficacy endpoint.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 96
logMAR | -0.0519 (0.0075)

2. Secondary Outcome: Mean Difference Between Achieved and Target Corneal Flap Thickness as Assessed by OCT
Description: The expected flap thickness as determined pre-operatively was subtracted from the achieved flap thickness as assessed by optical coherence tomography (OCT) (ie, an imaging method using light to capture three-dimensional images). A positive number represents a postoperative flap thickness that is thicker than the expected flap thickness and vice versa for a negative number.
Time Frame: Operation/Surgery (Day 1), Month 1 Postoperative, Month 6 Postoperative
Population: This analysis population includes all subjects with 1 month post-operative measurements of the primary efficacy endpoint with data at the specific time point.
Measure: Mean (Standard Deviation); unit: microns
Groups:
- Operation/Surgery (Day 1); Month 1 Postoperative; Month 6 Postoperative: WaveLight Refractive Suite
Arm/Group | Operation/Surgery (Day 1) | Month 1 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 96 | 96 | 95
microns
  Right Eye | 3.958 (11.0173) | 3.448 (7.6679) | 3.200 (7.0795)
  Left Eye | 3.905 (12.2162) | 3.427 (7.5096) | 2.253 (5.8854)

3. Secondary Outcome: Mean Manifest Refraction (Sphere)
Description: Manifest refraction was performed under photopic lighting conditions using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart at 4 meters. The subject was manually refracted to his/her best correction using a phoropter. Each eye individually contributed to the mean.
Time Frame: Baseline (Day 0), Operation/Surgery (Day 1), Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: Eyes
Groups:
- Baseline/Screening (Day 0); Day 1 Postoperative; Month 1 Postoperative; Month 3 Postoperative; Month 6 Postoperative: WaveLight Refractive Suite
Arm/Group | Baseline/Screening (Day 0) | Day 1 Postoperative | Month 1 Postoperative | Month 3 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 96 | 96 | 96 | 96 | 95
Number analyzed (Eyes) | 192 | 192 | 192 | 192 | 190
diopter | -3.672 (1.9820) | 0.046 (0.3318) | 0.077 (0.3474) | 0.046 (0.3426) | 0.017 (0.3383)

4. Secondary Outcome: Mean Manifest Refraction (Cylinder)
Description: Manifest refraction was performed under photopic lighting conditions using an ETDRS chart at 4 meters. The subject was manually refracted to his/her best correction using a phoropter. Each eye individually contributed to the mean.
Time Frame: Baseline (Day 0), Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: Eyes
Arm/Group | Baseline/Screening (Day 0) | Month 1 Postoperative | Month 3 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 96 | 96 | 96 | 95
Number analyzed (Eyes) | 192 | 192 | 192 | 190
diopter | -0.32 (0.860) | -0.16 (0.254) | -0.16 (0.217) | -0.18 (0.244)

5. Secondary Outcome: Mean Laser Treatment Time
Description: Treatment time with Excimer EX500 and Femtosecond FS200 lasers, measured in seconds.
Time Frame: Day 0 (surgery)
Population: This analysis group includes all participants with 1 month post-operative measurement of the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- EX500 Laser: Excimer 500 laser used during LASIK surgery for corneal ablation
- FS200 Laser: Femtosecond FS200 laser used during LASIK surgery for corneal ablation
Arm/Group | EX500 Laser | FS200 Laser
Number analyzed (Participants) | 96 | 96
seconds
  Right eye (OD) | 9.912 (3.5755) | 30.161 (19.1352)
  Left eye (OS) | 9.709 (3.4498) | 29.214 (16.4972)

6. Secondary Outcome: Mean Total Laser Treatment Time
Description: Total treatment time with Excimer EX500 and Femtosecond FS200 lasers, measured in seconds. Total duration for both eyes was calculated as sum of duration for the right eye and left eye.
Time Frame: Day 0 (surgery)
Population: This analysis group includes all participants with 1 month post-operative measurement of the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | WaveLight Refractive Suite
Number analyzed (Participants) | 96
seconds
  Right eye (OD) | 40.073 (19.1612)
  Left eye (OS) | 38.923 (16.6188)
  Both eyes | 78.996 (32.6967)

7. Secondary Outcome: Mean Response: "Rate Your Vision, Over the Past 4 Weeks, With NO Glasses or Contact Lenses"
Description: As recorded by the subject on the the Refractive Status and Vision Profile (RSVP), a self-reported questionnaire used to measure vision-related health status in persons with refractive error, on a scale from 0 (completely blind) to 10 (perfect vision).
Time Frame: Baseline (Day 0), Month 1 Postoperative, Month 6 Postoperative
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline (Day 0); Month 1 Postoperative; Month 6 Postoperative: WaveLight Refractive Suite
Arm/Group | Baseline (Day 0) | Month 1 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 80 | 95 | 94
units on a scale | 3.6 (1.71) | 9.1 (1.08) | 9.4 (0.78)

8. Secondary Outcome: Percent Response by Category: "In the Past 4 Weeks, to See Far Away, I Wore..."
Description: As recorded by the subject on the RSVP questionnaire, where n/a means no use of glasses or contact lenses.
Time Frame: Baseline (Day 0), Month 1 Postoperative, Month 6 Postoperative
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Baseline (Day 0) | Month 1 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 96 | 96 | 95
percentage of subjects
  only glasses | 36.5 | 1.0 | 0.0
  mostly glasses, sometimes contact lenses | 32.3 | 0.0 | 0.0
  about equally, glasses and contact lenses | 17.7 | 0.0 | 0.0
  mostly contact lenses, sometimes glasses | 11.5 | 0.0 | 0.0
  only contact lenses | 1.0 | 0.0 | 0.0
  n/a | 1.0 | 99.0 | 100.0

9. Secondary Outcome: Percent Response by Category: "I Worry About my Vision"
Description: As recorded by the subject on the RSVP questionnaire
Time Frame: Baseline (Day 0), Month 1 Postoperative, Month 6 Postoperative
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Baseline (Day 0) | Month 1 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 96 | 96 | 95
percentage of subjects
  Never | 10.4 | 21.9 | 52.6
  Rarely | 30.2 | 51.0 | 33.7
  Sometimes | 40.6 | 19.8 | 11.6
  Often | 13.5 | 7.3 | 2.1
  Always | 5.2 | 0.0 | 0.0

10. Secondary Outcome: Percent Response by Category: "My Vision Is a Concern in My Daily Life"
Description: As recorded by the subject on the RSVP questionnaire
Time Frame: Baseline (Day 0), Month 1 Postoperative, Month 6 Postoperative
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Baseline (Day 0) | Month 1 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 96 | 96 | 95
percentage of subjects
  Never | 6.3 | 27.1 | 63.2
  Rarely | 34.4 | 51.0 | 27.4
  Sometimes | 34.4 | 14.6 | 5.3
  Often | 14.6 | 5.2 | 3.2
  Always | 10.4 | 2.1 | 1.1

11. Secondary Outcome: Percent Response by Category: "Driving at Night"
Description: As recorded by the subject on the RSVP questionnaire, where 0 is "Not applicable", 1 is "No difficulty at all", 2 is "A little difficulty", 3 is "Moderate difficulty", 4 is "Severe difficulty" and 5 is "So much difficulty that I did not do the activity with this alternative".
Time Frame: Baseline (Day 0), Month 1 Postoperative, Month 6 Postoperative
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Baseline (Day 0) | Month 1 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 96 | 96 | 95
percentage of subjects
  With glasses, 0 | 4.2 | 100.0 | 100.0
  With glasses, 1 | 38.5 | 0.0 | 0.0
  With glasses, 2 | 34.4 | 0.0 | 0.0
  With glasses, 3 | 18.8 | 0.0 | 0.0
  With glasses, 4 | 4.2 | 0.0 | 0.0
  With glasses, 5 | 0.0 | 0.0 | 0.0
  With contact lenses, 0 | 38.5 | 100.0 | 100.0
  With contact lenses, 1 | 36.5 | 0.0 | 0.0
  With contact lenses, 2 | 20.8 | 0.0 | 0.0
  With contact lenses, 3 | 4.2 | 0.0 | 0.0
  With contact lenses, 4 | 0.0 | 0.0 | 0.0
  With contact lenses, 5 | 0.0 | 0.0 | 0.0
  Without glasses/contact lenses, 0 | 29.2 | 3.1 | 0.0
  Without glasses/contact lenses, 1 | 0.0 | 43.8 | 73.7
  Without glasses/contact lenses, 2 | 0.0 | 40.6 | 21.1
  Without glasses/contact lenses, 3 | 4.2 | 8.3 | 4.2
  Without glasses/contact lenses, 4 | 8.3 | 3.1 | 1.1
  Without glasses/contact lenses, 5 | 58.3 | 1.0 | 0.0

12. Secondary Outcome: Mean Contrast Sensitivity (CS)
Description: Contrast sensitivity (ie, the ability to detect slight changes in luminance before they become indistinguishable) was assessed binocularly with distance manifest correction in place and uncorrected. Contrast sensitivity was assessed at spatial frequencies of 3, 6, 12, and 18 cycles per degree (cpd), where 3.0 cpd = A, 6.0 cpd = B, 12.0 cpd = C, and 18.0 cpd = D. Raw scores were log transformed. A higher numeric value represents better contrast sensitivity.
Time Frame: Baseline (Day 0), Day 1 Postoperative, Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative
Population: This analysis population includes all subjects with 1 month post-operative measurements of the primary efficacy endpoint. Here, "n" is the number of subjects assessed uncorrected.
Measure: Mean (Standard Deviation); unit: logCS
Arm/Group | Baseline (Day 0) | Day 1 Postoperative | Month 1 Postoperative | Month 3 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 96 | 96 | 96 | 96 | 95
logCS
  CS A (uncorrected), n=84, 84, 90, 96, 95 | 0.768 (0.4356) | 1.845 (0.1340) | 1.868 (0.1433) | 1.894 (0.1168) | 1.898 (0.1311)
  CS B (uncorrected), n=84, 84, 90, 96, 95 | 0.937 (0.3991) | 2.035 (0.1650) | 2.096 (0.1341) | 2.134 (0.1267) | 2.117 (0.1354)
  CS C (uncorrected), n=84, 84, 90, 96, 95 | 0.623 (0.3995) | 1.734 (0.2065) | 1.806 (0.1734) | 1.835 (0.1640) | 1.854 (0.1485)
  CS D (uncorrected), n=84, 84, 90, 96, 95 | 0.189 (0.4188) | 1.273 (0.2059) | 1.378 (0.1773) | 1.401 (0.1517) | 1.411 (0.1380)
  CS A (corrected) | 1.808 (0.1399) | 1.863 (0.1485) | 1.900 (0.1300) | 1.922 (0.1242) | 1.917 (0.1327)
  CS B (corrected) | 2.020 (0.1880) | 2.056 (0.1631) | 2.116 (0.1352) | 2.151 (0.1217) | 2.148 (0.1265)
  CS C (corrected) | 1.739 (0.2095) | 1.757 (0.1925) | 1.828 (0.1517) | 1.857 (0.1391) | 1.876 (0.1441)
  CS D (corrected) | 1.281 (0.2014) | 1.311 (0.2025) | 1.402 (0.1577) | 1.427 (0.1346) | 1.432 (0.1299)

13. Secondary Outcome: Wavefront Aberrometry
Description: Wavefront aberrations (optical imperfections of the eye that prevent light from focusing perfectly on the retina, resulting in defects in the visual image) were measured using a commercially available system. Higher order aberrations (i.e., spherical aberrations, coma, and trifoil) are defined as optical imperfections which cannot be corrected by any reliable means of present technology.
Time Frame: Baseline (Day 0), Month 6 Postoperative
Population: This analysis population includes all subjects with 1 month post-operative measurements of the primary efficacy endpoint.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Baseline (Day 0) | Month 6 Postoperative
Number analyzed (Participants) | 96 | 95
microns
  Total Higher Order RMS, Right Eye | 0.7 (0.97) | 0.5 (0.42)
  Total Higher Order RMS, Left Eye | 0.7 (1.12) | 0.5 (0.42)
  Spherical Aberrations, Right Eye | 0.1 (0.27) | 0.2 (0.13)
  Spherical Aberrations, Left Eye | 0.1 (0.19) | 0.2 (0.17)
  Coma, Right Eye | 0.3 (0.42) | 0.3 (0.27)
  Coma, Left Eye | 0.3 (0.43) | 0.3 (0.19)
  Trifoil, Right Eye | 0.3 (1.02) | 0.4 (0.61)
  Trifoil, Left Eye | 0.3 (0.79) | 0.3 (0.57)

14. Secondary Outcome: Corneal Curvature as Measured by Keratometry
Description: Corneal curvature was assessed by a commercially available system and measured in diopters.
Time Frame: Baseline (Day 0), Month 1 Postoperative, Month 3 Postoperative, Month 6 Postoperative
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: diopter
Arm/Group | Baseline (Day 0) | Month 1 Postoperative | Month 3 Postoperative | Month 6 Postoperative
Number analyzed (Participants) | 96 | 96 | 96 | 95
diopter
  K1, Right Eye | 43.5 (1.41) | 40.4 (1.79) | 40.6 (1.76) | 40.6 (1.76)
  K1, Left Eye | 43.5 (1.46) | 40.4 (1.89) | 40.5 (1.88) | 40.5 (1.83)
  K2, Right Eye | 43.9 (1.55) | 40.8 (1.91) | 41.0 (1.91) | 41.0 (1.87)
  K2, Left Eye | 44.0 (1.57) | 40.8 (1.97) | 40.9 (1.96) | 41.0 (1.93)
  Mean K1 and K2, Right Eye | 43.7 (1.38) | 40.6 (1.81) | 40.8 (1.79) | 40.8 (1.77)
  Mean K1 and K2, Left Eye | 43.8 (1.42) | 40.6 (1.90) | 40.7 (1.89) | 40.7 (1.84)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of the study (23 Sep 2013 through 12 Aug 2014). This analysis group includes all enrolled participants.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the medical device.
Groups:
- WaveLight Refractive Suite: Excimer EX500 and Femtosecond FS200 lasers (Wavelight® Refractive Suite) used during LASIK surgery for corneal flap creation and corneal ablation
- Screen Failure: Prior to treatment
Arm/Group | WaveLight Refractive Suite | Screen Failure
Serious Adverse Events (participants affected / at risk) | 1/97 | 0/7
Other Adverse Events (participants affected / at risk) | 0/97 | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | WaveLight Refractive Suite (N=97) | Screen Failure (N=7)
Cerebrovascular accident (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.